CLINICAL TRIAL: NCT05282420
Title: Ranibizumab Versus Aflibercept for Macular Edema Secondary to Non-ischemic Central Retinal Vein Occlusion in Young Adult Patients.
Brief Title: Ranibizumab Versus Aflibercept for CRVO in Young Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Ahmed Amer, Ophthalmology department Qena Faculty of medicine, South Valley University, Egypt, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU\MED\Oph026\4\21\12\284
Record Dates: First submitted 2022-03-04; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Non-Ischemic Central Retinal Vein Occlusion With Macular Edema
Keywords: non ischemic CRVO; Macular edema; Ranibizumab; Aflibercept
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two groups, twenty patients (20 eyes) each. The first group received 0.5 mg\0.1 ml ranibizumab intravitreal injections and the second group received 2.0 mg\0.1 ml aflibercept intravitreal injections. all patients were followed up for at least 12 months.
  Patients were given the planned treatment throughout the study and no switching was done between anti-VEGF drugs
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ranibizumab group (Active Comparator): Ranibizumab injection monthly for 3 successive months
  Interventions: Procedure: intravitreal injection of Ranibizumab; Drug: Ranibizumab
- Aflibercept group (Active Comparator): Aflibercept injection monthly for 3 successive months
  Interventions: Procedure: intravitreal injection of Aflipercept; Drug: Aflibercept

INTERVENTIONS:
Procedure: intravitreal injection of Ranibizumab — intravitreal injection of Anti-VEGF Ranibizumab (Lucentis®; manufactured in the United States by Genentech/Roche)
  Arms: Ranibizumab group
Procedure: intravitreal injection of Aflipercept — intravitreal injection of Anti-VEGF Aflibercept (Eylea®; manufactured in the United States)
  Arms: Aflibercept group
Drug: Ranibizumab — Ranibizumab
  Arms: Ranibizumab group
Drug: Aflibercept — Aflipercept
  Arms: Aflibercept group

SUMMARY:
this study will compare the efficacy and safety of use either Ranibizumab and Aflibercept in treatment of macular edema resulting from non ischemic central retinal vein occlusion in patients younger than 5o years old

DETAILED DESCRIPTION:
This is a prospective randomized interventional study, Forty eyes of forty patients younger than 50 years with macular edema due to non-ischemic CRVO were enrolled in the study.

Patients will be randomized into 2 groups. First group will receive intravitreal injection of Ranibizumab 0.5 mg\0.1ml. the second group will receive intravitreal injection of 2.0 mg\0.1 ml Aflibercept. All patients will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients younger than 50 years with macular edema due to non-ischemic CRVO

Exclusion Criteria: Other conditions that might affect the macula as

1. diabetic retinopathy, intraocular inflammation, age related macular degeneration, patients with solar or radiation retinopathy,
2. patients with ischemic type CRVO and patients who had recent intraocular surgery.
3. patients who had previous intravitreal injections, ophthalmic laser surgeries.
4. patients with dense cataracts whom fundus was difficult to scan.
5. Patients who were lost to follow up visits were also excluded

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity BCVA | at 12 months post-injection
  change BCVA after injection

SECONDARY OUTCOMES:
reduction of macular edema | at 12 months post-injection
  change in central subfield macular thickness CST on OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Ali Ahmed Amer, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes